CLINICAL TRIAL: NCT06473233
Title: Interest of TEG6S® in Reducing Transfusion Needs During Postpartum Haemorrhage
Acronym: INTEGRAL-HPP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0013
Record Dates: First submitted 2024-06-12; First posted 2024-06-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Before TEG6S: Patients managed in a period of 12 months before the implementation of TEG6S®
- After TEG6S: Patients managed in a period of 12 months after the implementation of TEG6S®
  Interventions: Device: TEG6S

INTERVENTIONS:
Device: TEG6S — Hemostatic management including one or more delocalized biology test with the TEG6S®, at the discretion of the responsible clinician
  Groups: After TEG6S

SUMMARY:
The main objective of this study is to evaluate fibrinogen consumption, transfusion need, and other security outcomes in women with postpartum hemorrhage of 1000 mL or more, before and after the implementation of a TEG6S® device at a level III maternity unit (Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France).

DETAILED DESCRIPTION:
Acquired obstetrical coagulopathy during massive postpartum hemorrhage (PPH) is a serious and frequent complication of delivery. It has been shown that fibrinogen levels are the first to fall during PPH, and that a level inferior to a threshold of 2g/L is strongly associated with progression to severe PPH, hemostatic impairment, transfusion, and invasive hemostatic procedures.

The clinical diagnosis of coagulopathy is difficult, and the biological diagnosis by usual laboratory tests is often delayed, leading to the empirical administration of fibrinogen and blood products, sometimes unnecessary.

The TEG6S® is a viscoelastic testing device performed on whole blood, which allows a reliable assessment of hemostasis and coagulation quality in about ten minutes.

The anomalies detected by the TEG6S® allow for the early diagnosis of acquired coagulopathy, especially hypofibrinogenemia. Its use during the management of PPH would therefore allow for transfusion savings and potential economic benefits, in addition to improving patient prognosis through early and appropriate treatment (including the absence of early "blind" treatment in the absence of coagulopathy).

ELIGIBILITY:
Inclusion Criteria:

* Woman of 18 years old or more
* Delivery at the level III maternity of Centre Hospitalier Sud Francilien (CHSF) (Corbeil-Essonnes, France) between 2022 and 2024, except deliveries during cyber-attack period at CHSF (from August 2022 to December 2022 included), due to uncertainty over the completeness of the data.
* Presenting postpartum hemorrhage with estimated blood loss of 1000mL or more
* No constitutional hemostasis anomaly
* No treatment interfering with hemostasis
* No use of blood products and/or pro-coagulant products before delivery

Exclusion Criteria:

- Patient informed of the research and refusing the use of the data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women who gave birth at the level III maternity of Centre Hospitalier Sud Francilien and had postpartum haemorrhage greater than 1000mL or more.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Fibrinogen consumption | up to 24 hours
  Quantity of fibrinogen administered (in grams)

SECONDARY OUTCOMES:
Total number of TEG6S® | at 12 months
  Total number of TEG6S® carried out over a period of 12 months following its implementation
Estimated blood loss | up to 24 hours
  Estimated total volume of blood loss during PPH, in milliliters, using a graduated bag and weight of blood-soaked materials
Calculated blood loss | up to 24 hours
  Estimated total volume of blood loss during PPH, using the following formula = ([initial Ht - Ht H24] × total blood volume × 100/35) + compensated blood loss (CBL) ; with: total blood volume in milliliters = basis weight × 65 × 1.4, and CBL in milliliters, corresponding to the number of RBC concentrates transfused (1 RBC corresponds to approximately 500 mL of blood at 35% Ht).
Consumption of packed red blood cells (RBC) | up to 24 hours
  Number of packed red blood cells used
Consumption of fresh frozen plasma (FFP) | up to 24 hours
  Number of fresh frozen plasma (FFP) used
Invasive haemostatic procedure | up to 24 hours
  Use of surgical and/or radio-interventional hemostasis (Bakri balloon, embolization, arterial ligation, uterine padding, hemostasis hysterectomy)
Maternal death | until leaving the hospital
  Occurrence of maternal death at hospital
ICU admission | until leaving the hospital
  Any admission in an intensive care unit
ICU length of stay | until discharge from the intensive care unit
  Total length of stay in an intensive care unit/critical care (in days)
Total length of stay | until discharge from the intensive care unit
  Total length of stay in hospital (in days)
Acute anemia | at 24 hours
  Occurrence of anemia following postpartum hemorrhage, defined by a decrease in hemoglobin level of 4g/dL or more at 24h following delivery, compared to the last hemoglobin level known before delivery

CONTACTS AND LOCATIONS:
Overall Officials: Fatima BRIK, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No